CLINICAL TRIAL: NCT02206698
Title: Multicenter, Prospective Development of a Clinical Prediction Model to Determine Which Children Can Safely Avoid Abdominal CT Scanning During the Initial Evaluation of Blunt Abdominal Trauma
Brief Title: Pediatric Blunt Abdominal Trauma Clinical Prediction Model
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: Monroe Carell Jr. Children's Hospital at Vanderbilt (Other); University of Arkansas (Other); University of Alabama at Birmingham (Other); Virginia Commonwealth University (Other); Children's Mercy Hospital Kansas City (Other); University of Tennessee (Other); Memorial Hermann Hospital (Other); Baylor College of Medicine (Other); Children's Hospital Los Angeles (Other); Children's Hospital Medical Center, Cincinnati (Other); Washington University School of Medicine (Other); Boston Children's Hospital (Other); Emory University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00030071
Record Dates: First submitted 2014-07-31; First posted 2014-08-01 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Pediatric Abdominal Trauma
Keywords: Intraabdominal Injury; CT Abdomen and Pelvis; Pediatric trauma; blunt abdominal injury; blunt trauma; clinical prediction model
MeSH Terms: conditions — Wounds, Nonpenetrating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The submitted proposal is designed to reduce morbidity and mortality to injured children. Significant variability in the initial trauma assessment exists among institutions. The proposed project is a prospective, observational, multi-institutional study of children following blunt abdominal trauma. The specific goals of the project are to: 1) Document history, physical exam findings, imaging, and laboratory values, which are available to physicians during the initial trauma resuscitation prior to a decision on whether to order an abdominal computed tomography (CT) to evaluate for potential intra-abdominal injury; and 2) Derive and validate a multi-variable clinical prediction rule based on data variables readily available during the pediatric trauma resuscitation to identify patients at low risk for intra-abdominal injury, in which unnecessary CT might safely be avoided. Information from this study could be used to develop a more standardized approach to the evaluation for intra-abdominal injury following blunt trauma in children. This information could lead to significant improvement in the early recognition of injury and to improved resource utilization.

DETAILED DESCRIPTION:
The proposed research project is a prospective, observational study. Data will be collected from each institution and entered into a secure REDCap database. Two phases of data collection will occur: 1) patient demographics and specific clinical variables which may be associated with IAI which are available and recorded during the initial trauma evaluation 2) laboratory and imaging results available after the initial assessment, identified injuries, patient disposition, interventions and outcomes.

Primary Outcome Variables: 1) Intra-abdominal injury (IAI) (presence of solid or hollow organ injury (spleen, liver, kidney, GI tract, adrenal, pancreas, intra-abdominal vascular structure, bladder, ureter, gallbladder, abdominal wall fascia)) 2) IAI requiring intervention (abdominal operation, angio-embolization, blood transfusion)

Time Course: The initial data collection period will extend for one year. Data will be recorded in a password protected redcap database which is readily available online to all participating institutions.

Study setting: Eleven Level One Pediatric Trauma Centers

Data collection points: demographics (age, mechanism, alert level), physical exam, labs (AST, HCT, amylase, UA, base deficit), FAST, imaging results, injuries, outcomes (admission, ICU admit, need for intervention, missed injuries, ISS).

Data Analysis: De-identified data will be used during the data analysis phase to minimize the risk of loss of confidentiality to the patients. Data analysis with development of a clinical prediction rule (CPM) will be performed as follows. A logistic regression will be used to fit a predictive model for both IAI and IAI requiring interventions. SAS 9.3 will be used for the statistical analysis. Validation (including sensitivity and negative predictive value) of the derived CPM would then be performed in a subsequent study using a second population of patients. Internal validation of the prediction model was assessed by creating a split sample using a random selection process; half of the sample was used as the initial cohort to develop the prediction model for estimates of all covariates, and the remaining half was used as the validation cohort to compare the true to the predicted outcomes. A receiver operating characteristic (ROC) curve is created by plotting sensitivity against (1- specificity) for different cut-off points of the predicted outcome. A bootstrap study of 1000 replications was performed on the level of sensitivity, specificity and TP/FP/FN/TN validation. Validation (including sensitivity and negative predictive value) of the derived CPM would then be performed in a subsequent study using a second population of patients.

Quality assurance plan: Data quality will be evaluated bi-monthly by a team consisting of the PI, an expert in clinical prediction models and a statistician. This panel will be able to review de-identified data from all institutions but will not have access to make any changes in the data entered in the centralized database.

Data checks to compare data entered into the registry against predefined rules for range or consistency: Data checks to compare entered registry data against predefined rules for range and consistency will be performed bi-monthly.

Source data verification: Source data collection is the responsibility of each individual institution. A data analysis team consisting of a statistician and an expert in clinical prediction models will evaluate the data bi-monthly to look for wide outliers (beyond pre-defined range) and impossible data values (not clinically possible) and request clarification from the individual institutions when necessary.

Data dictionary that contains detailed descriptions of each variable: The vast majority of the data collection points are discrete variables with no opportunity for "free text" data entry. Many of these variables are specifically described on the data collection tools. Data definitions and question from the individual sites are addressed in a frequently updated Frequently Asked Questions (FAQ) document which is sent out to the sites bi-monthly following data verification review.

Standard Operating Procedures to address registry operations and analysis activities: The database is established through a secure Vanderbilt Redcap web-based site. Individual site data collection will be analyzed and reviewed bi-monthly with feedback to each of the sites if data inconsistencies exist.

Plan for missing data to address situations where variables are reported as missing, unavailable, "non-reported," cannot be interpreted, or considered missing because of data inconsistency or out-of-range results: Critical data which are missing, unavailable or not reported will not be utilized for the development of the blunt abdominal trauma clinical prediction model (BAT CPM). The investigators will attempt clarification for out of range results prior to data analysis. Variables which are available and reported in less than 50% of the patients will likely be excluded from the CPM because they will not form the basis of a practicable risk stratification model. The developed CPM will require validation in a second un-related population prior to widespread application of the CPM.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting as a Trauma system activation with suspicion for blunt abdominal trauma. (Fall >10 feet; Motor vehicle accident >40mph, pedestrian struck by auto, Motor vehicle crash with ejection or death in vehicle or rollover, assault, bicycle accident, ATV accident).
* <16 years of age
* The need to activate the trauma system is dictated by the Emergency Department physician
* Consults called to the department of surgery for suspicion of intraabdominal traumatic injury

Exclusion Criteria:

* 16 years of age or older
* Burn injury
* Hanging
* Drowning
* Penetrating injury
* CT A/P performed prior to arrival
* Presentation >6 hours from time of injury
* Pregnancy
* Isolated head injury
* Fall <10 feet with no concern for intraabdominal injury
* Isolated extremity injury

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with blunt abdominal trauma
Sampling Method: Non-Probability Sample
Enrollment: 2800 (Actual)
Dates: Start 2014-07; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Intra-abdominal Injury (IAI) | 30 days from time of trauma
  Intra-abdominal injury (IAI) (presence of solid or hollow organ injury (spleen, liver, kidney, GI tract, adrenal, pancreas, intra-abdominal vascular structure, bladder, ureter, gallbladder, abdominal wall fascia))
Intraabdominal Injury (IAI) requiring intervention | 30 days from time of trauma
  Intra-abdominal injury (IAI) requiring intervention (Laparoscopy or Laparotomy, angio-embolization, blood transfusion for IAI)

CONTACTS AND LOCATIONS:
Overall Officials: Christian J Streck, MD, Principal Investigator — Medical University of South Carolina
Locations (14):
- United States (14):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - LA Children's, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - Boston Children's, Boston, Massachusetts
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Le Bonheur Children's Hospital, The University of Tennessee Health Science Center, Memphis, Tennessee
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Children's Hospital of Richmond, Richmond, Virginia

REFERENCES:
- [Derived] Frederick AB, Vogel AM, Williams RF, Zhang J, Huang EY, Savoie KB, Santore MT, Tsao K, Falcone RA, Dassinger MS, Haynes JH, Russell RT, Naik-Mathuria BJ, St Peter SD, Mooney DP, Onwubiko C, Blakely ML, Streck CJ. Multicenter external validation of the Pediatric Emergency Care Applied Research Network rule to identify children at very low risk for intra-abdominal injury requiring acute intervention. J Trauma Acute Care Surg. 2025 Jun 1;98(6):966-972. doi: 10.1097/TA.0000000000004597. Epub 2025 Apr 2. PMID 40170217